CLINICAL TRIAL: NCT07319403
Title: Comparison of the Effects of Hip and Ankle Focused Progressive Exercise Training on Lower Extremity Function in Athletes With Chronic Ankle Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Çiğdem Demir, Student, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU-FTR-ÇD-01
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Ankle Sprains
Keywords: Ankle Injuries; Muscle Strength; Exercise Training
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Participants with chronic ankle instability will be randomly assigned into three parallel groups: a gluteus medius strengthening group, a gluteus maximus strengthening group, and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gluteus Maximus (Experimental): Participants with chronic ankle instability will participate in a 6-week hip-focused exercise program emphasizing gluteus maximus activation.
  Interventions: Other: Gluteus Maximus
- Gluteus Medius (Experimental): Participants with chronic ankle instability will participate in a 6-week hip-focused exercise program emphasizing gluteus medius activation.
  Interventions: Other: Gluteus Medius
- Control (Active Comparator): Participants with chronic ankle instability will participate in a 6-week exercise program commonly used in the rehabilitation of ankle instability
  Interventions: Other: Control

INTERVENTIONS:
Other: Gluteus Medius — Participants with chronic ankle instability will undergo a 6-week hip-focused strengthening exercise program specifically targeting the gluteus medius muscle. The intervention aims to improve hip muscle strength and lower extremity stability.
  Arms: Gluteus Medius
Other: Gluteus Maximus — Participants with chronic ankle instability will participate in a 6-week hip-focused strengthening exercise program targeting the gluteus maximus muscle. The program aims to enhance hip extension strength and overall lower extremity stability.
  Arms: Gluteus Maximus
Other: Control — Participants with chronic ankle instability will perform a 6-week standard strengthening exercise program commonly used in the rehabilitation of ankle instability, without specific emphasis on targeted hip muscle strengthening.
  Arms: Control

SUMMARY:
Chronic ankle instability refers to a combination of persistent mechanical and functional instability symptoms following an ankle sprain. Along with these symptoms, decreased proprioception, reduced neuromuscular control, poor postural control, limited dorsiflexion range of motion, decreased ankle strength, and altered lower-extremity biomechanics during functional activities are also observed. In addition, individuals with chronic ankle instability have been shown to exhibit limitations in energy transfer across the lower extremity. These symptoms may hinder patients' physical activity levels and athletic performance and negatively affect their quality of life. Since the lower extremity functions as a unit, changes in adaptive strategies at the ankle can lead to kinematic alterations in proximal joints. Although the instability originates at the ankle, higher-level joints are also affected, and it has even been reported that in this population, lower-extremity stability is primarily achieved through the hip joint. While the effectiveness of hip-focused exercises has begun to be investigated in the literature, the superiority of different muscle groups has not yet been compared.

DETAILED DESCRIPTION:
Chronic ankle instability is characterized by persistent mechanical and functional impairments that may develop following a lateral ankle sprain. Individuals with this condition commonly exhibit reduced proprioception, impaired neuromuscular control, limited dorsiflexion range of motion, and altered lower-extremity biomechanics, all of which may negatively affect daily activities and athletic performance. These deficits often lead to compensatory strategies at more proximal segments, and emerging evidence suggests that hip musculature plays a meaningful role in maintaining dynamic ankle stability. However, the specific contribution of individual hip muscle groups has not yet been clearly defined.

This study is designed to compare the effects of strengthening different hip muscle groups -the gluteus medius and gluteus maximus- on functional and neuromuscular outcomes in individuals with chronic ankle instability. Participants will be randomly assigned to one of three parallel groups: a gluteus medius strengthening group, a gluteus maximus strengthening group, or a control group performing standard balance exercises. Each intervention group will follow a structured and progressively loaded exercise program targeting the designated muscle group. All participants will complete supervised training sessions throughout the intervention period.

The study protocol includes a baseline assessment session, a multi-week intervention phase, and a post-intervention evaluation. Outcome measures will include functional performance tests, assessments of neuromuscular control, and metrics related to dynamic stability. These outcomes will be collected before and after the intervention to determine differences between groups.

The aim of this protocol is to determine whether targeted strengthening of specific hip muscle groups yields superior improvements in individuals with chronic ankle instability. The findings are expected to enhance understanding of the role of proximal musculature in lower-extremity stability and contribute to more precise and effective rehabilitation strategies for this population.

ELIGIBILITY:
Inclusion Criteria:

Professional athletes aged between 18 and 40 years

Participation in sports for at least 3 years

History of at least one lateral ankle sprain that occurred at least 12 months prior to enrollment

At least two episodes of perceived ankle "giving way" and/or at least two recurrent lateral ankle sprains within the past 6 months, and/or a subjective feeling of ankle instability on the injured side

Exclusion Criteria:

History of lower extremity surgery

History of fracture involving the lower extremity

Any lower extremity injury within the past 3 months that limited physical activity for more than one day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool (CAIT) | Baseline and after 6 weeks
  The Cumberland Ankle Instability Tool (CAIT) is a self-reported questionnaire designed to assess the severity of chronic ankle instability. It consists of 9 items evaluating ankle stability during daily and sports-related activities. Scores range from 0 to 30, with lower scores indicating greater perceived ankle instability. An increase in the CAIT score reflects clinical improvement in ankle stability.

SECONDARY OUTCOMES:
Functional Ankle Instability Questionnaire | Baseline and after 6 weeks
  Self-reported functional ankle instability will be evaluated using the Functional Ankle Instability Questionnaire. The questionnaire will be administered face-to-face by a trained physiotherapist to assess perceived ankle instability during daily and sports-related activities.
Hip Muscle Strength | Baseline and after 6 weeks
  Isometric hip abduction and hip extension muscle strength will be assessed using a handheld dynamometer (KForce Muscle Controller, KInvent, USA). Hip abduction strength will be measured in a side-lying position at 25° of hip abduction with the knee extended, targeting the gluteus medius muscle. Hip extension strength will be measured in a prone position with the knee flexed at 90°, targeting the gluteus maximus muscle. Three trials will be performed bilaterally, and the mean value will be used for analysis.
Side Hop Test | Baseline and after 6 weeks
  Functional performance will be assessed using the Side Hop Test. Participants will be instructed to perform repeated lateral hops on one leg over a single reference line as quickly as possible for 30 seconds. The total number of successful hops will be recorded. The test will be performed three times, and the highest value will be used for analysis.
Step-Down Test | Baseline and after 6 weeks
  Postural stability and lower extremity kinematics will be evaluated using the Step-Down Test. Participants will stand on a raised platform on the test limb with hands placed on the waist and perform a controlled step-down by lowering the contralateral heel toward the ground and returning to the starting position. The movement will be performed at a standardized pace. The movement quality will be evaluated based on trunk, pelvis, and knee alignment.
Y-Balance Test | Baseline and after 6 weeks
  Dynamic balance will be assessed using the Y-Balance Test. Participants will perform maximal reach distances in the anterior, posteromedial, and posterolateral directions while standing on the dominant limb. Reach distances will be normalized to limb length. The average of three trials in each direction will be used for analysis.
Single-Leg Heel Raise Balance Test | Baseline and after 6 weeks
  Static balance will be assessed using the single-leg heel raise balance test. Participants will stand on one leg and perform plantar flexion while maintaining balance. The test will be terminated when the heel touches the ground. The average duration of three trials will be recorded.
Weight-Bearing Lunge Test | Baseline and after 6 weeks
  Ankle dorsiflexion range of motion will be assessed using the weight-bearing lunge test. Participants will lunge forward toward a wall while maintaining heel contact with the ground. The maximum distance between the great toe and the wall will be measured. Three trials will be performed for each limb, and the mean value will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Düzgün, Principal Investigator — Hacettepe University; Gülcan Harput, Principal Investigator — Ankara Medipol University
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Law on the Protection of Personal Data (LPPD)